CLINICAL TRIAL: NCT01263353
Title: An Open-label Phase I Study Evaluating the Safety and Tolerability of Pasireotide LAR in Combination With Everolimus in Advanced Metastatic NETs - The COOPERATE-1 Study
Brief Title: Safety and Tolerability of Pasireotide LAR in Combination With Everolimus in Advanced Metastatic NETs
Acronym: COOPERATE-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSOM230F2102; 2010-018895-26 (EudraCT Number)
Record Dates: First submitted 2010-12-16; First posted 2010-12-20 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2016-04

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumor of the Pulmonary ot Gastroenteropancreatic System
Keywords: Carcinoid tumor,; Gastroenteropancreatic Neuroendocrine Tumors,; Pulmonary Neuroendocrine Tumors,; pasireotide LAR,; SOM230 LAR,; everolimus,; RAD001,; Advanced Neuroendocrine Tumor,; Gastroenteropancreatic System
MeSH Terms: conditions — Carcinoid Tumor | interventions — Everolimus

ARMS (6):
- Functional tumors, pre-treated (Experimental)
  Interventions: Drug: Pasireotide LAR followed by Pasireotide LAR + Everolimus
- Functional tumors, treatment naïve (Experimental)
  Interventions: Drug: Pasireotide LAR followed by Pasireotide LAR + Everolimus
- Nonfunctional tumors, pretreated 1 (Experimental)
  Interventions: Drug: Pasireotide LAR followed by Pasireotide LAR + Everolimus
- Nonfunctional tumors, pretreated 2 (Experimental)
  Interventions: Drug: Everolimus followed by Pasireotide LAR + Everolimus
- Nonfunctional tumors, treatment-naïve 1 (Experimental)
  Interventions: Drug: Pasireotide LAR followed by Pasireotide LAR + Everolimus
- Nonfunctional tumors, treatment-naïve 2 (Experimental)
  Interventions: Drug: Everolimus followed by Pasireotide LAR + Everolimus

INTERVENTIONS:
Drug: Pasireotide LAR followed by Pasireotide LAR + Everolimus
  Arms: Functional tumors, pre-treated; Functional tumors, treatment naïve; Nonfunctional tumors, pretreated 1; Nonfunctional tumors, treatment-naïve 1
Drug: Everolimus followed by Pasireotide LAR + Everolimus
  Arms: Nonfunctional tumors, pretreated 2; Nonfunctional tumors, treatment-naïve 2

SUMMARY:
The purpose of this study is to assess the safety and tolerability of pasireotide LAR in combination with everolimus in advanced metastatic gastroenteropancreatic or pulmonary neuroendocrine Tumors (NET).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of grade 1/2 advanced pulmonary or gastroenteropancreatic neuroendocrine tumor
* Progressive disease within last 12 months (only patients with nonfunctional tumors)
* Documented liver metastasis
* Measurable disease per RECIST determined by multiphase MRI or triphasic CT

Exclusion Criteria:

* Previous treatment with radiolabeled somatostatin analogs within 12 months prior to reporting baseline symptoms
* Previous treatment with mTOR inhibitors or pasireotide
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study
* Women who are pregnant or lactating

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Evaluate safety and tolerability profile of pasireotide LAR in combination with everolimus in patients with advanced metastatic NET | 3 months

SECONDARY OUTCOMES:
Evaluate safety and tolerability of pasireotide LAR and/or everolimus in patients with advanced metastatic NET | 15 months
To assess pharmacokinetic exposures of pasireotide LAR and everolimus during monotherapy and in combination therapy | 15 months
To assess potential drug-drug interactions between pasireotide and everolimus during combination therapy | 12 months
To assess symptom control (bowel movements and flushing episodes) with pasireotide LAR in combination with everolimus in patients with functioning tumors | 15 months
To assess the biochemical response (chromograninA, CgA) to pasireotide LAR in combination with everolimus | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Germany (4):
  - Novartis Investigative Site, Bad Berka
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Münster

REFERENCES:
- See also: Results for CSOM230F2102 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13569